CLINICAL TRIAL: NCT05594927
Title: A Prospective, Randomized, Parallel-Controlled, Double-Blind, Double-Dummy, Multicenter, Phase III Clinical Trial of Icaritin Soft Capsule Versus Huachansu Tablet in the First-line Treatment of Unresectable Hepatocellular Carcinoma With Poor Conditions and Biomarker Enrichment (Biomarker Enrichment Study of Poor Prognosis HCC Patients, BESTPOP)
Brief Title: Icaritin Soft Capsule Versus Huachansu Tablet in the First-line Treatment of Unresectable Hepatocellular Carcinoma With Poor Conditions and Biomarker Enrichment (Biomarker Enrichment Study of Poor Prognosis HCC Patients, BESTPOP)
Acronym: BESTPOP
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing Shenogen Biomedical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SNG2111-ICR-1
Record Dates: First submitted 2022-10-17; First posted 2022-10-26 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Hepatocellular Carcinoma
Keywords: Icaritin, Poor Conditions, Composite Biomarker; First-line Treatment
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — icaritin; huachansu

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Icaritin soft capsule (Experimental)
  Interventions: Drug: Icaritin
- Huachansu tablet (Active Comparator)
  Interventions: Drug: Huachansu

INTERVENTIONS:
Drug: Icaritin — 600 mg (6 x 100 mg capsules) icaritin administered orally twice daily (30 minutes after breakfast and dinner, respectively) until treatment discontinuation criteria are met.
  Arms: Icaritin soft capsule
Drug: Huachansu — 1200 mg (4 x 300 mg tablets) huachansu administered orally three times a day (30 minutes after breakfast, lunch and dinner, respectively) until treatment discontinuation criteria are met.
  Arms: Huachansu tablet

SUMMARY:
A study to evaluate the efficacy and safety of icaritin versus huachansu in the first-line treatment of unresectable hepatocellular carcinoma with poor conditions and biomarker enrichment.

DETAILED DESCRIPTION:
This is a prospective, randomized, parallel-controlled, double-blind, double-dummy, multicenter, phase III clinical trial. Patients with poor conditions and biomarker enrichment will be randomly assigned in a 2:1 ratio to receive either icaritin or huachansu as the first-line treatment until unacceptable toxic effects and loss of clinical benefit. A total of 261 participants with 206 deaths are required. The primary endpoint is overall survival (OS) in the full analysis set (FAS) population.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18 years and older;
2. HCC patients who meet the clinical diagnostic criteria of the Chinese Diagnosis and Treatment Guideline of Primary Liver Cancer (2022 edition), and/or with diagnosis confirmed histopathologically/cytologically;
3. Unresectable HCC patients;
4. Patients with a peripheral blood composite biomarker Score ≥ 2 points, 1 point each for AFP ≥ 400 ng/mL, TNF-α < 2.5 pg/mL, and IFN-γ ≥ 7.0 pg/mL ;
5. No prior first-line systemic treatment for HCC, including sorafenib, lenvatinib, donafenib, atezolizumab plus bevacizumab, sintilimab plus a bevacizumab biosimilar, camrelizumab plus apatinib, and durvalumab plus tremelimumab, oxaliplatin-based systemic chemotherapy (FOLFOX4) , icaritin, huachansu, and other anti-cancer drugs such as targeted agents, immune checkpoint inhibitors, and systemic chemotherapy;
6. Child-Pugh score ≤ 7;
7. Vital organ functions should meet the following requirements:

   ① Hematopoietic function: platelet ≥ 40×10^9/L, hemoglobin ≥ 80 g/L, white blood cell ≥ 2.0×10^9/L;

   ② Liver function: total bilirubin ≤ 1.5 times upper limit of normal (ULN) , alanine Aminotransferase (ALT) and aspartate Aminotransferase (AST) ≤ 5×ULN; albumin ≥ 28 g/L;

   ③ Renal function: Serum Creatinine ≤ 1.5×ULN, or creatinine clearance rate ≥ 50 mL/min;
8. If HBV-DNA ≥ 10^4 copies/mL (2000 IU/mL), antiviral and liver protection therapy must be used before enrollment, until HBV-DNA < 10^4 copies/mL (2000 IU/mL). In which case, the antiviral drugs should be administered continuously and liver function and hepatitis B virus load will be monitored during the study period;
9. Patients who meet one of two conditions: (A) are not or less appropriate candidates for first-line standard treatments recommended by the guidelines; (B) are not willing to receive first-line standard treatments recommended by the guidelines.
10. Surgical resection ended > 3 months, local ablation, hepatic artery intervention or radiotherapy ended > 4 weeks before randomization (implantation of radioactive particles ended > 3 months) and relevant adverse reactions having recovered. Patients without extrahepatic spread must have radiographic evidence of disease progression after local treatment;
11. Patients who had previously received adjuvant systemic therapy after surgical resection experienced the first radiographic disease progression more than 6 months after withdrawal of adjuvant therapy will be eligible for enrollment;
12. Within 2 weeks prior to randomization, no treatment with modern Chinese traditional medicine preparations with anti-tumor indications (refer to the 11th inclusion criterion when huaier granule was used as systemic adjuvant therapy), immunomodulators such as interferon-α and thymalfasin, tumor vaccines and cellular immunotherapy;
13. No blood transfusion or infusion of blood products, no use of hematopoietic growth factors (such as granulocyte colony-stimulating factor G-CSF), and no albumin infusion within 2 weeks prior to randomization;
14. ≥1 measurable lesion according to the Response Evaluation Criteria In Solid Tumors (RECIST 1.1), defined as a non-lymphoid lesion with the longest diameter ≥ 10 mm or a lymph node lesion with the short axis ≥ 15 mm; a lesion after previous radiotherapy or other loco-regional therapy which has been demonstrated progression confirmed per RECIST v1.1 with the longest diameter ≥ 10 mm scanned by dynamic-enhanced CT/ dynamic-enhanced MRI is to be deemed as a measurable lesion.
15. Eastern Cooperative Oncology Group (ECOG) performance score (PS) of 0 or 1;
16. Expected survival of ≥ 12 weeks;
17. Female patients of childbearing age with a negative blood pregnancy within the first 7 days prior to randomization will be eligible; Female patients of childbearing age or male patients with female sexual partners of childbearing age should take effective contraceptive measures throughout treatment and within 3 months after the last dose;
18. Voluntary agreement to sign informed consent and the willingness and ability to comply with protocol schedules and testing;
19. No treatment with any other investigational drugs or medical devices within 4 weeks prior to randomization.

Exclusion Criteria:

1. Tumor occupancy ≥ 70% of liver, or tumor thrombus occupancy ≥ 50% of the main trunk of portal vein, or mesenteric vein or inferior vena cava tumor thrombus;
2. Moderate-to-severe ascites, i.e., the score of the indicator is > 2; Moderate-to-severe, or symptomatic pleural effusion and pericardial effusion requiring drainage;
3. Receipt of major surgery (craniotomy, thoracotomy, laparotomy, hip replacement, etc.) within 28 days prior to randomization or planned to receive major surgery during the study;
4. Other types of primary liver cancer, such as intrahepatic cholangiocarcinoma, mixed HCC and cholangiocarcinoma, fibrolamellar HCC, etc. Other malignancies within 5 years prior to signing the informed consent form or at present, excluding radically treated basal cell carcinoma of skin, squamous cell carcinoma of skin and/or radically resected carcinoma in situ;
5. Pregnant or lactating women;
6. Grade 2 or above myocardial ischemia or myocardial infarction (NCI-CTCAE v5.0), poorly-controlled arrhythmia, and/or New York Heart Association (NYHA) class III or IV cardiac insufficiency;
7. Patients who previously received allogeneic transplantation including liver transplantation, or plan to undergo liver transplantation during the study;
8. History of hepatic encephalopathy and/or hepatic nephropathy within 6 months prior to signing informed consent ;
9. HCV-RNA positive, ALT and/or AST > 2×ULN;
10. Human immunodeficiency virus (HIV) antibody positive;
11. Severe infection (≥ Grade 3 of NCI-CTCAE v5.0 criteria) at randomization;
12. Unable to swallow, chronic diarrhea or intestinal obstruction, which will significantly affect oral administration and absorption of the study drug;
13. History of gastrointestinal hemorrhage within 6 months before signing informed consent, or with clear tendency for gastrointestinal hemorrhage at present, such as: local active ulcers, stool occult blood ≥ 2+ or positive at two consecutive tests (attention should be paid to exclude the influence of food, drugs and other diseases);
14. Active autoimmune diseases requiring systemic treatment (e.g., NSAIDs, immunosuppressants, biologics, corticosteroids, etc.) except for patients receiving replacement therapy (e.g., hypothyroidism treated with thyroxine, type 1 diabetes mellitus treated with insulin, adrenal or pituitary insufficiency treated with physiologic corticosteroids, etc.);
15. Known central nervous system (CNS) metastasis; patients suspected of CNS metastasis need to undergo cerebral MRI/CT for exclusion;
16. Significant coagulation function abnormalities: international standardized ratio (INR) > 1.5 or prothrombin time (PT) > 16 s;
17. History of schizophrenia or psychiatric drug abuse;
18. Known allergy or intolerance to any ingredients of icaritin or huachansu preparations;
19. Other conditions that the investigator considers inappropriate for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 261 (Estimated)
Dates: Start 2022-12-12 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | From randomization to death from any cause, assessed up to approximately 24 months
  Defined as the time from randomization to death from any cause

SECONDARY OUTCOMES:
9/12/18-month overall survival (OS) rate | From randomization to 9, 12 and 18 months later
  Defined as the percentage of participants who are alive at 9, 12, 18 months following randomization
Time to progression (TTP) | From randomization to the first occurrence of disease progression, assessed up to approximately 24 months
  Defined as the time from randomization to the first occurrence of disease progression, as determined by the investigator and IRC according to RECIST v1.1
Progression--free survival (PFS) | From randomization to the first occurrence of disease progression or death from any cause (whichever occurs first), assessed up to approximately 24 months
  Defined as the time from randomization to the first occurrence of disease progression or death from any cause (whichever occurs first), as determined by the investigator and IRC according to RECIST v1.1
Objective response rate (ORR) | Up to approximately 24 months after randomization
  Defined as the percentage of participants with complete response (CR) or partial response (PR), as determined by the investigator and IRC according to RECIST v1.1
Disease control rate (DCR) | Up to approximately 24 months after randomization
  Defined as the percentage of participants with complete response (CR), partial response (PR) or stable disease (SD), as determined by the investigator and IRC according to RECIST v1.1
Time to deterioration (TTD) | From randomization to first deterioration, assessed up to approximately 24 months
  Defined as the time from randomization to first deterioration, i.e., decrease or increase from baseline of ≥ 10 points in the following EORTC QLQ-C30 and EORTC QLQ-HCC18 subscales respectively, maintained for two consecutive assessments or one assessment followed by death from any cause within 4 weeks:
Adverse events (AEs) | Up to approximately 24 months after randomization
  Defined as all untoward medical events in a participant administered the study drug, which can be symptoms, signs, diseases or laboratory abnormalities, irrespective of the causality with the study drug.
  The type, incidence, severity, and relationship with study drugs of adverse events (AEs) will be evaluated.
Trough plasma concentration (Cmin） | Pre-dose at the end of cycle1 (Cycle length=28 days)
  Defined as trough plasma concentration（Cmin）of icaritin and its metabolites
Maximum plasma concentration (Cmax) | Post-dose at the end of cycle1 (Cycle length=28 days)
  Defined as maximum plasma concentration (Cmax) of icaritin and its metabolites
Mean area under the concentration-time curve during the dosing interval (AUC0-t) | Within 0.5 h before dosing (0 h) and 0.5 h, 1 h, 2 h, 3 h, 4 h, 6 h, 8 h, 10 h, and 12 h after dosing at the end of cycle1 (Cycle length=28 days)
  Defined as Mean area under the concentration-time curve during the dosing interval (AUC0-t) of icaritin and its metabolites at steady state

CONTACTS AND LOCATIONS:
Overall Officials: Jihui Hao, MD, Principal Investigator — Tianjin Medical University Cancer Institute and Hospital
Locations (3):
- China (3):
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Chifeng Municipal Hospital, Chifeng, Mongolia
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No